CLINICAL TRIAL: NCT04976478
Title: A Perspective, Multi-center, Single Arm Study of Nimotuzumab Combined With IMRT in Elder Patients With Cervical Squamous Cell Carcinoma
Brief Title: Study of Nimotuzumab Combined With IMRT in Elder Patients With Cervical Squamous Cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Junjie Wang, Department director, Peking University Third Hospital
Other Study IDs: ChiECRCT20210238
Record Dates: First submitted 2021-07-02; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Cervical Squamous Cell Carcinoma
MeSH Terms: interventions — nimotuzumab; Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: All patients will be treated with Nimotuzumab combined with radiotherapy.
  Interventions: Drug: Nimotuzumab; Radiation: EBRT combined with brachytherapy

INTERVENTIONS:
Drug: Nimotuzumab — Patients receive Nimotuzumab: 200mg, intravenous infusion, weekly for 6 weeks.
Radiation: EBRT combined with brachytherapy — IMRT/VMAT are adopted. A total dose of 45-50.4 Gy, 1.8~2.0Gy/f, 25~ 28F in pelvic and/or extension filed. For patients with metastasis in pelvic lymph node and abdominal para-aortic lymph node, the dose of radiation in local lesion will be increased to 60~66Gy. For patients at stage IIIB, concurrent radiation will be given in parametrial extension or in the late course the dose will be increased to 60Gy.
  Brachytherapy: Three dimensional high dose rate brachytherapy is used with HR-CTV D90 cumulative dose of 80~85Gy (EQD2); If the tumor diameter is ≥4cm, HR-CTV D90 cumulative dose is ≥87Gy (EQD2). Brachytherapy combined with external beam radiotherapy will be completed within 8 weeks.

SUMMARY:
To evaluate the efficacy and safety of Nimotuzumab combined with IMRT in elder patients with locally advanced cervical squamous cell carcinoma

DETAILED DESCRIPTION:
This is a perspective, multi-center, open-label and single arm study.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥65 years old
2. Histologically confirmed primary cervical squamous cell carcinoma in stage IB3-IVA (FIGO 2018)
3. At least one measurable lesion according to RECIST 1.1 guideline
4. Patients are intolerant to or refuse chemotherapy.
5. No serious hematopoietic dysfunction, nor abnormal heart, lung, liver and kidney function, nor immunity deficiency. And the results of lab test meet the following criteria:

   Hemoglobin ≥90g/L Absolute count of neutrophils≥2×109/L orwhite blood cell count≥4.0×109/L； Platelet count≥100×109/L； AST≤2.5×ULN ALT≤2.5×ULN TBIL≤1.5×ULN；

   Serum creatinine≤1.5×ULN or CrCl> 60 mL/min(according toCockcroft-Gault):

   Serum creatinine≤1.5×ULN Female CrCl=(140-Age)×Weight（kg）×0.85 / (72×Scr mg/dl)
6. ECOG score 0-2
7. Expectancy of life is at least 3 months.
8. Eligible for pelvic MRI examination.
9. The patients voluntarily received nimotuzumab combined with radiotherapy.
10. Patients can comply with the protocol and are willing to sign informed consent.

Exclusion Criteria:

1. Patients who have received treatment for cervical cancer, including surgery, radiotherapy, chemotherapy, targeted therapy and immunotherapy
2. Patients who have bilateral ureteral obstruction, who cannot be placed ureteral stents or perform pyelostomy.
3. Patients with rectovaginal fistula/vaginovesical fistula/uncontrolled vaginal bleeding or with fistula risk.

.4)Patients infected with HIV. 5)Active hepatitis B (HBV DNA quantitative test results exceed the detection threshold), or HCV infection (HCV RNA quantitative test results exceed the detection threshold) 6)Patients with severe underlying disease that makes it possible to safely receive the treatment. And the severe underlying disease include but not limited to active infections requiring systemic medication, decompensated heart failure (NYHA grade III and IV), unstable angina pectoris, and acute myocardial infarction occurred within the first 3 months of enrollment.

7)Patients with a history of prior malignancy other than cured basal cell carcinoma of the skin.

8)Patients with Crohn's disease and ulcerative colitis. 9)Patients are allergic to Nimotuzumab or its compounds. 10)Patients with neurological or psychiatric abnormalities that affect cognitive ability.

11)Intracavitary brachytherapy cannot be performed that was assessed by the investigator.

12)Other factors were assessed by investigators to be unsuitable to this study.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The elder patients with cervical squamous cell cancer received nimotuzumab combined with radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival(DFS) | up to 3 years
  The rate of patient without disease in 3 years after treatment

SECONDARY OUTCOMES:
Complete response rate(CRR) | 3 months later after treatment
  The percentage of subjects who achieve complete response by imaging assessment from the end of the treatment to disease progression
Objective response rate(ORR) | 3 months later treatment
  The percentage of patients who experienced complete or partial cancer shrinkage or disappearance after treatment
3-year overall survival(OS) | up to 3 years
  The rate of patient alive in 3 years after treatment
The change of tumor related markers | up to 3 years
  the correlation of the value of SCC，Cyfra 21-1 and therapeutic effect [The changes of serum tumor markers (such as SCC-Ag and CYFRA21-1) were observed before and after treatment]
The change of cervical tumor | At diagnosis and before brachytherapy
  the change of the volume of the cervical tumor at diagnosis and before brachytherapy
QUALITY OF LIFE(QoL) | up to 3 years
  Quality of life assessed by EORTC QLQ-CX 24 [EORTC QLQ-CX 24 is a specific quality of life assessment scale based on EORTC QLQ-C 30, with 24 items]
SAFETY | up to 3 years
  Including severity of adverse events, the incidence of adverse events and serious adverse events. Adverse events should be reported and graded according to CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No